CLINICAL TRIAL: NCT03310970
Title: Absolute Bioavailability/Pharmacokinetic and Residual Drug Analysis of Topical Lidocaine in Healthy Adults
Brief Title: Pharmacokinetics of Lidocaine in Healthy Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nicole K Brogden (Other)
Collaborators: Long Island University (Other)
Responsible Party: Sponsor-Investigator, Nicole K Brogden, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 201701725
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Results first posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Healthy
Keywords: Peer Reviewed Research
MeSH Terms: interventions — Lidocaine; Transdermal Patch; Lidoderm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lidocaine 5% patch (Active Comparator): Each subject will wear three generic Lidocaine 5% topical patches for 12 hours.
  Interventions: Drug: Lidocaine 5% patch
- Lidoderm® 5% patch (Active Comparator): Each subject will wear three Lidoderm® topical patches for 12 hours.
  Interventions: Drug: Lidoderm 5% patch
- Intravenous lidocaine (Active Comparator): A single intravenous dose of 0.5 mg/kg lidocaine hydrochloride will be administered to each subject.
  Interventions: Drug: Lidocaine hydrochloride

INTERVENTIONS:
Drug: Lidocaine 5% patch — Each subject will wear three generic Lidocaine 5% topical patches for 12 hours.
  Arms: Lidocaine 5% patch
Drug: Lidocaine hydrochloride — Each subject will receive a dose of 0.5 mg/kg intravenously over a period of 5 minutes.
  Arms: Intravenous lidocaine
Drug: Lidoderm 5% patch — Each subject will wear three Lidoderm® topical patches for 12 hours.
  Arms: Lidoderm® 5% patch

SUMMARY:
The study to be performed will utilize already FDA-approved marketed products in healthy adults for the purpose to generate data for establishing rate of drug delivery of Lidoderm® topical patch (manufactured by Endo Pharmaceuticals) and the lidocaine 5% patch (manufactured by Mylan Pharmaceuticals) in healthy adults, and to ensure the safety of individuals utilizing these types of products.

DETAILED DESCRIPTION:
Topical drug delivery systems in the form of patches are convenient, attractive, and easy to use. Lidocaine is a very popular patch available on the United States market today. Accurate determination of the rate and extent of drug release and absorption is crucial to ensure the safety of individuals using these and other types of patches. The drug delivery rate can be determined early in the development process by using in vitro skin flux permeation studies, and later in humans by accurately quantifying residual drug from patches post-wear and in pharmacokinetic studies. In this study the investigators will employ two types of evaluation to determine the rate and extent of drug release and absorption from lidocaine patches, namely residual drug analysis post-wear and pharmacokinetic analysis in healthy adult volunteers. In addition, the investigators will compare the serum drug concentrations following patch and intravenous administration in order to determine the absolute bioavailability of these patches. Positive outcomes of this project will identify appropriate methods to determine the rate and extent of drug release and absorption from topical patches, and will help regulatory agencies in the development of Guidances for Industry regarding the characterization of drug release and absorption kinetics to ensure the safety of individuals utilizing these types of products.

ELIGIBILITY:
Inclusion Criteria:

1. Men or non-pregnant women, of any ethnic background, between the age of 18 and 65 years old.
2. Provide written informed consent before initiation of any study procedures.
3. Available for follow-up for the planned duration of the study.
4. Able to communicate well with the investigators.
5. Demonstrate comprehension of the protocol procedures and knowledge of study, as demonstrated by a study member filling out a consent checklist form to verify that the subject understands all aspects of the study including the purpose, procedures, risks and benefits.
6. Able to adhere to the study protocol schedule, study restrictions and examination schedule.
7. Subjects must be non-smokers and not regular users of tobacco. They must have refrained from regular and habitual use of nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, gum, patch or electronic cigarettes) over the previous 12 months and must have not used any nicotine-containing products in the previous 30 days.
8. Subjects who are within their ideal body weight (BMI between 18-29.9 kg/m2).
9. Subjects deemed to be healthy as judged by the Medically Accountable Investigator (MAI), as determined by medical history, physical examination, and medication history.
10. Negative urine drug screening test.
11. Have a normal blood pressure (systolic: 90-139 mmHg; diastolic: 60-89 mmHg) and heart rate (55-100 bpm).
12. Have normal screening laboratories for WBC, Hgb, Hct, platelets, sodium, potassium, chloride, bicarbonate, BUN, creatinine, ALT, AST.
13. Female subjects must be of non-childbearing potential. This is defined as surgically sterile (i.e. history of hysterectomy or tubal ligation), or postmenopausal for more than 1 year (no bleeding for 12 consecutive months). If the person is of childbearing potential they must be non-pregnant at the time of enrollment and on the morning of the first day of each study treatment procedure day (a urine pregnancy test will be administered if it has been >30 days since serum pregnancy test for enrollment). The person must also agree to use hormonal or barrier birth control such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner.
14. Agrees not to participate in another clinical study during the study period unless the study is in the follow-up phase and it has been one month since the subject received any experimental agents or treatments. The subject also agrees not to participate in an investigational drug study for at least 30 days after last procedure day.
15. Agrees not to donate blood to a blood bank throughout participation in the study and for at least 60 days after last procedure day.
16. Have a normal ECG; must not have any of the following: pathologic Q wave abnormalities, significant ST-T wave changes, left ventricular hypertrophy, right bundle branch block, left bundle branch block, advanced A-V heart block, non-sinus rhythm, excluding isolated premature atrial contractions (sinus rhythm is not between 55-100 beats per minute), or any other abnormality that, in the opinion of the MAI, makes it unsafe for the subject to participate in the study.

Exclusion Criteria:

1. Women who are pregnant or lactating or have a positive serum pregnancy test at enrollment or positive urine pregnancy test at any time during the study.
2. Smokers. A "smoker", for the purposes of the study, will be defined as an individual who has regularly and habitually used nicotine-containing substances, including tobacco products (e.g., cigarettes, cigars, chewing tobacco, gum, patch or electronic cigarettes) over the past 12 months. Occasional recreational use (less than once monthly) will not warrant exclusion unless the individual has used nicotine-containing substances in the previous 30 days before study enrollment.
3. Participation in any ongoing investigational drug trial or clinical drug trial period unless the study is in the follow-up phase and it has been ≥ one month since the subject received any experimental agents or treatments.
4. Abnormal vital signs, defined as:

   * Hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg) at rest on two separate days.
   * Heart rate <55 at rest on two separate days
   * Respiratory rate ≤ 11 to ≥ 18 breaths per minute
5. Temperature >38.0ºC (100.4ºF) or symptoms of an acute self-limited illness such as an upper respiratory infection or gastroenteritis within seven days of administration of a study product.
6. History of chronic obstructive pulmonary disease.
7. Positive urine drug screening test.
8. Use of any prescription medication during the period 0 to 30 days or over-the counter medication during the period 0 to 3 days before entry to the study (vitamins, herbal supplements and birth control medications will be allowed).
9. Use of medications or treatments that would significantly influence or exaggerate responses to the test product or that would alter inflammatory or immune response to the product. This includes antihistamines (within 72 hours prior to dosing), systemic or topical corticosteroids within four weeks prior to dosing, use of monoamine oxidase inhibitors 21 days prior to study, cyclosporine, tacrolimus, cytotoxic drugs, immune globulin, Bacillus Calmette-Guerin [BCG], monoclonal antibodies, or radiation therapy.
10. Donation or loss of greater than one pint of blood within 60 days of entry to the study.
11. Any prior serious adverse reaction or hypersensitivity to lidocaine administered by any route.
12. Current diagnosis of any major psychiatric illness.
13. Received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 30 days before enrollment in this study or expects to receive an experimental agent during the study.
14. Medical history of a serious chronic condition, including (but not limited to): allergic conditions such as anaphylaxis to food or drugs; asthma; generalized drug reactions; any seizure disorder; any central nervous system disorder; glaucoma (open or closed angle); history of pyloric or urinary bladder neck obstruction; intestinal obstruction; difficulty swallowing; stomach or bowel problems (e.g, blockage, muscle weakness, ulcerative colitis, Crohn's disease); bleeding disorders; acid reflux disease; myasthenia gravis; allergy to belladonna alkaloids; impaired hepatic or renal function.
15. Any condition that would, in the opinion of the Principal Investigator (PI) or MAI, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
16. Inability to communicate or cooperate with the investigators.
17. Medical history of significant dermatologic diseases or conditions, such as atopy, psoriasis, vitiligo or conditions known to alter skin appearance or physiologic response (e.g. diabetes, porphyria).
18. History of significant dermatologic cancers (e.g. melanoma, squamous cell carcinoma), except basal cell carcinomas that were superficial and did not involve the investigative site.
19. History of consumption of alcohol within 24 hours prior to dose administration.
20. Subject has an obvious difference in skin color at patch sites (compared to neighboring skin), or the presence of a skin condition, excessive hair at the application site, sunburn, raised moles and scars, open sores at application site, scar tissue, tattoo, or coloration that would interfere with placement of test articles, or the assessment of the skin and/or reactions to drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-10-09 (Actual); Study Completion 2019-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole K Brogden, PharmD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at the University of Iowa by advertisements in the "Noon News", a UIHC newsletter, and by a mass email that was sent to all staff/faculty/and students. Recruitment began in March 2018 and continued until the enrollment goal was reached in October 2019.
Groups:
- Group 1: Generic Lidocaine Patches First, IV Lidocaine Second, the Lidoderm(R) Topical Patches Last: Each subject in this group received study interventions in the following order:
  Each subject first wore three generic 5% (Mylan Pharmaceuticals, 140mg) lidocaine patches for 12 hours, followed by a minimum washout period of 24 hours. Each subject then received a single intravenous dose of 0.5 mg/kg lidocaine hydrochloride, followed by a minimum washout period of 24 hours. Each subject then wore three lidoderm(R) 5% (Endo Pharmaceuticals, 700mg) lidocaine patches for 12 hours.
- Group 2: Lidoderm(R) Topical Patches First, IV Lidocaine Second, Then Generic Lidocaine Patches Last: Each subject in this group received study interventions in the following order:
  Each subject first wore three lidoderm(R) 5% (Endo Pharmaceuticals, 700mg) lidocaine patches for 12 hours, followed by a minimum washout period of 24 hours. Each subject then received a single intravenous dose of 0.5 mg/kg lidocaine hydrochloride, followed by a minimum washout period of 24 hours. Each subject then wore three generic 5% (Mylan Pharmaceuticals, 140mg) lidocaine patches for 12 hours.
Period: Overall Study
Arm/Group | Group 1: Generic Lidocaine Patches First, IV Lidocaine Second, the Lidoderm(R) Topical Patches Last | Group 2: Lidoderm(R) Topical Patches First, IV Lidocaine Second, Then Generic Lidocaine Patches Last
Started | 11 | 12
Completed | 11 | 11
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Measure Description: Analysis of all study participants that received all three interventions as well as the 1 subject who withdrew consent prior to completing all study procedures.
Groups:
- All Study Participants: All study participants received IV lidocaine, generic lidocaine patches, and Lidoderm patches.
Arm/Group | All Study Participants
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.9 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 20
  Asian | 2
  Hispanic/Latino | 1
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 23.7 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Maximum Serum Concentration of Lidocaine (Cmax)
Description: Cmax is the highest lidocaine concentration measured in the serum.
Time Frame: For both patch arms measured at time points: 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 24, 27, 30, 33, 36, 39, 48 hours. For intravenous lidocaine hydrochloride arm measured at time points: 2, 5, 10, 20, 30, 45 minutes, 1, 2, 3, 4, 6, 8, 10 hours.
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- All Study Participants: All subjects analyzed received and completed the following interventions:
  Each of the subjects wore three lidocaine 5% (Mylan Pharmaceuticals) patches for 12 hours.
  Each of the subjects wore three lidoderm® 5% (Endo Pharmaceuticals) topical patches for 12 hours.
  Each of the subjects received a single intravenous 0.5 mg/kg dose of lidocaine hydrochloride.
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
ng/ml
  Lidocaine 5% patch | 113.95 (38.84)
  Lidoderm® 5% patch | 123.54 (68.97)
  Intravenous lidocaine hydrochloride | 706.15 (338.86)

2. Secondary Outcome: Measurement of Volume of Lidocaine Distribution (V)
Description: Volume of distribution is a mathematical concept that relates the amount of lidocaine in the body to the concentration of lidocaine measured in the serum.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/kg
Groups:
- All Study Participants: Each subject received all of the following interventions:
  Each subject wore three generic 5% (Mylan Pharmaceuticals) lidocaine patches for 12 hours.
  Each subject wore three lidoderm(R) 5% (Endo Pharmaceuticals) lidocaine patches for 12 hours.
  Each subject received a single intravenous dose of 0.5 mg/kg lidocaine hydrochloride.
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
L/kg
  Lidocaine 5% patch | 5.13 (2.07)
  Lidoderm® 5% patch | 5.15 (2.13)
  Intravenous lidocaine hydrochloride | 1.98 (0.68)

3. Secondary Outcome: Measurement of Time of Maximum Serum Lidocaine Concentration (Tmax).
Description: Tmax is the time point at which the maximum drug concentration in serum is measured.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
hours
  Lidocaine 5% patch | 9.08 (2.90)
  Lidoderm® 5% patch | 10.82 (2.2)
  Intravenous lidocaine hydrochloride | 0.03 (0)

4. Secondary Outcome: Measurement of Elimination Rate Constant of Lidocaine (Kel)
Description: The elimination rate constant is a mathematical value describing the rate at which lidocaine is removed from the body.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
1/hr
  Lidocaine 5% patch | 0.17 (0.06)
  Lidoderm® 5% patch | 0.19 (0.12)
  Intravenous lidocaine hydrochloride | 0.31 (0.1)

5. Secondary Outcome: Determination of Area Under the Serum-concentration-time Curve (AUC)
Description: Area under the serum-concentration-time curve is a mathematical measure of total systemic exposure to lidocaine in the body.
Time Frame: For both patch arms measured at time points: 1, 2, 3, 4, 5, 6, 8, 10, 12 hours. For intravenous lidocaine hydrochloride arm measured at time points: 2, 5, 10, 20, 30, 45 minutes, 1, 2, 3, 4, 6, 8, 10 hours.
Measure: Mean (Standard Deviation); unit: ng*h/ml
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
ng*h/ml
  Lidocaine 5% patch | 807.32 (285.31)
  Lidoderm® 5% patch | 748.55 (420.93)
  Intravenous lidocaine hydrochloride | 671.07 (165.01)

6. Secondary Outcome: Residual Drug Analysis in Worn TDDS and Patches
Description: The amount of drug remaining in the patches is measured after the patches have been worn and removed. This outcome is only reported for the patch arms of the study and is not applicable to the intravenous arm.
Time Frame: Measured after patches are removed from subjects following 12 hours of patch wear.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
mg
  Lidocaine 5% patch | 123.79 (6.58)
  Lidoderm® 5% patch | 655.16 (29.96)

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from the date of consent, during study intervention and washout (12 days), and for 2 days of follow-up after study procedures were completed (14 days total).
Description: Adverse Events were collected based on subject reporting of events. While not all 23 participants were included in the data assessment, Adverse events were recorded for all 23 study participants. While all participants completed all three arms of the study, 1 participant withdrew after completing the Intravenous Lidocaine and Lidoderm Topical Patch Arm, leaving only 22 participants to be analyzed in the lidocaine patch arm.
Groups:
- Lidocaine Patch: Each subject will wear three generic lidocaine patches for 12 hours.
- Lidoderm ® Topical Patch: Each subject will wear three Lidoderm® topical patches for 12 hours.
Arm/Group | Lidocaine Patch | Lidoderm ® Topical Patch | Intravenous Lidocaine
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 19/22 | 19/23 | 17/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine Patch (N=22) | Lidoderm ® Topical Patch (N=23) | Intravenous Lidocaine (N=23)
Headache (General disorders) | 1 (1) | 2 (5) | 2 (5) — Participant reported
Increased Respiratory Rate (Respiratory, thoracic and mediastinal disorders) | 15 (34) | 13 (21) | 13 (50) — Respiratory Rate Normal Range: 12 - 17 breaths per minutes. Measured by nursing staff.
Increased Heart Rate (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (5) | 1 (1) — Heart Rate Normal Range: 55 - 100 beats per minutes. Measured by nursing staff
Decreased Heart Rate (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 8 (16) | 3 (5) — Heart Rate Normal Range: 55 - 100 beats per minute. Measured by nursing staff
Itchy lower back after patch removal (General disorders) | 1 (1) | 0 (0) | 0 (0) — Participant reported
Decreased Blood Pressure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) — Blood Pressure Normal Range: systolic (90-139 mmHg) diastolic (60-89 mmHg). Blood Pressure was recorded as decreased if either the systolic or diastolic was below normal range defined. Measured by nursing staff.
Increased Blood Pressure (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 2 (3) | 3 (3) — Blood Pressure Normal Range: systolic (90-139 mmHg) diastolic (60-89 mmHg). Blood Pressure was recorded as elevated if either the systolic or diastolic was above normal range defined. Measured by nursing staff
Lightheadedness (General disorders) | 0 (0) | 1 (1) | 1 (1) — Participant reported
Abnormal Hearing (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) — Any hearing changes reported by subjects (which were temporary and resolved prior to study end). For example, muffled hearing, ringing in the ears
Drowsiness/Sleepiness (General disorders) | 0 (0) | 0 (0) | 1 (1) — Patient reported
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Patient reported
Heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Participant reported
Contact erythema from IV placement (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Participant reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/70/NCT03310970/Prot_SAP_000.pdf